CLINICAL TRIAL: NCT04692883
Title: A Prospective Randomized Comparison of Functional Bracing Versus Rigid Immobilization After Modified Percutaneous Achilles Tendon Repair Under Local Anesthesia
Brief Title: Comparison of Functional Bracing vs Rigid Immobilization After Modified Percutaneous Achilles Tendon Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Maribor (Other)
Responsible Party: Principal Investigator, Andrej Cretnik, MD, PhD, principal investigator (Ass. Prof.), University Medical Centre Maribor
Other Study IDs: KME 54/03/00
Record Dates: First submitted 2020-12-22; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Achilles Tendon Rupture; Percutaneous Repair; Local Anesthesia; Postoperative Complications
Keywords: Achilles tendon; Percutaneous repair; Local anesthesia; Functional treatment; Early mobilization; Rigid immobilization
MeSH Terms: conditions — Postoperative Complications

INTERVENTIONS:
Procedure: Percutaneous suturing
  Other Names: Functional bracing

SUMMARY:
Rationale There is ongoing controversy over the optimal treatment and rehabilitation strategy of an acute Achilles tendon rupture (ATR). The highest general complication rate is reported in patients treated with percutaneous repair and early mobilization.

Objectives The purpose of the study is to compare the results of two ways of postoperative regimen after treatment with the modified and biomechanically significantly stronger percutaneous repair under local anesthesia.

Methods & Population All the consecutive patients with an acute complete Achilles tendon rupture who will agree to take part in a study will be randomized after a modified percutaneous repair under local anesthesia into functional group (FG), using a modified brace and immobilization group (IG), wearing a rigid plaster, in both groups for the period of 6 weeks. After that they will follow the same (standardized) rehabilitation protocol. Major and minor complication rate, diameter of the healed tendon, active and passive ankle range of motion (using neutral zero method), standing heel-rise test (with 25 repetition within a minute for a grade of normal) and clinical outcome using American Foot and Ankle Society (AOFAS) hindfoot-ankle score, return to the previous activity level, presence of associated complaints and subjective assessment (scored as good, fair or poor) will be assessed.

Time frame This will be a 4-year study with a 3-year follow-up.

Expected outcomes: There will be no differences in demographic parameters (age, gender, side and mechanism of the injury) between groups. Patients in the FG will reach sooner final range of motion (ROM) and muscular strength without limping and will be (subjectively) more satisfied with the treatment. There will be no statistically significant differences observed between groups according to the number of complications and in the end functional results with return to pre-injury activities.

DETAILED DESCRIPTION:
Rationale & background information There is ongoing controversy over the optimal treatment and rehabilitation strategy of an acute Achilles tendon rupture. Percutaneous suturing seems to bridge the gap between open surgical and conservative treatment, but still raises scepticism due to concerns like strength of the repair, approximation of torn ends, re-rupture rate, sural nerve injuries, early functional rehabilitation and thus final outcome. The highest general complication rate (15.6%) is reported in patients treated with percutaneous repair and early mobilization. The purpose of the study is to analyze the results of two ways of postoperative regimen after treatment with the modified and biomechanically significantly stronger percutaneous repair under local anesthesia.

Study goals and objectives The goals of the study are to compare the results of two ways of postoperative regimen after treatment with the modified and biomechanically significantly stronger percutaneous repair under local anesthesia . Objectives are to find whether the modified repair is strong enough to be used with functional treatment that enables more comfort and earlier rehabilitation to the patients with comparable end (functional) results and no more complications (particularly re-ruptures).

Study design

This will be a 4-year prospective observational study, with a 3-year follow up of all the consecutive patients who will meet the inclusion criteria:

1) patients 18 years of age or older; 2) a rupture that occurred no more than 7 days before the operating procedure; 3) closed, complete ATR; 4) a rupture that occurred in the tendinous portion (2-8 cm proximal to the insertion); 5) no previous operative procedures or history of partial or complete rupture of the involved tendon; 6) no previous local, oral or parenteral therapy that might have weakened the tendon (for instance local infiltration of anesthetics or steroids in the AT region, oral or parenteral immunosuppressive therapy in patients with transplanted organs or immune diseases etc.). The diagnosis must be confirmed clinically with palpable gap in the tendon, positive Thompson's test and inability of the patients to raise on their toes or heel. The diagnosis will be routinely checked by ultrasonography and in any case of doubt with MRI.

Methodology All the patients who agree to take part in a study will undersign informed/consent and will be operated on with the modified and biomechanically significantly stronger percutaneous repair under local anesthesia . After that they will be randomized after modified percutaneous suturing under local anesthesia in two groups - based on the day of Team A on service in the functional bracing group (FG) or based on the day of Team B in the group who will wear rigid immobilization (IG).

The first schedule will be on the second day (dressing), when functional brace or rigid immobilization will be applied in 25° of plantar flexion (PF). After that regular follow up will be after 3 and 6 weeks. In FG immobilization remains the same for 6 weeks, in IG it will be changed after 3 weeks and the foot put into neutral position. Patients in both groups will use crutches for assistance, and careful weightbearing of 5 to 10 kg will be allowed within first 3 weeks. Patients will be allowed to perform ROM exercises as much as their immobilization allows. After 3 weeks, patients may start with weightbearing as much as tolerated (until pain is felt).

After 6 weeks, all immobilization will be removed and patients in both groups will start with the rehabilitation according to the protocol (learned with physiotherapists). They are allowed to walk without crutches, with progressively increasing weightbearing (till tolerable pain) and ROM exercises with careful increasing of dorsiflexion (DF) (till 8 weeks in the sitting position and if possible, in water). Stretching exercises and squats with lifted heel will be allowed after 8 weeks (with a hand support between two chairs or tables and careful increasing of the load until pain is felt). Raising on toes or heels with the operated leg only will be allowed 12 weeks after the operation. Limited sports activities will be individually allowed after three months with recommended full loading 6 months after operation.

Major and minor complication rate, diameter of the healed tendon, active and passive ankle range of motion (using neutral zero method), standing heel-rise test (after 3 and 6 months if no pain is felt) and clinical outcome using AOFAS score will be observed. Return to the previous activity level, presence of associated complaints and subjective assessment (scored as good, fair or poor) will be also assessed. The outcome will be checked again after 1 and finally after 3 years. All the data will be recorded in the medical record (in computer), additional (manual) list is recorded with the investigators. Statistical analysis (parametric and non-parametric tests) will be performed (null hypothesis is that there will be no significant differences between the groups in the number of complications, particularly re-ruptures and in final results (type I and type II errors will be considered, p value less than 0.05 will be considered as statistically significant). In any case of complications patients can be scheduled anytime to the clinics in order to solve the problems.

Safety considerations Any patient can withdraw the study anytime - it has to be stated but in the medical record.

All the safety protocols must be respected and no harm produced to patients.

Follow-up Clinical follow-up will take part 3 years. Patients will be scheduled after 3 and 6 weeks and then after 2, 3 and 6 months and then after 1 and 3 years after the procedure.

Quality assurance The trial will follow the principles of good clinical practice - patients will be able to come to the clinics anytime if any complications occur and to withdraw the study at any time. All the data through will be recorded in the hospital data system and in the checking list of investigators and followed by the investigators and other clinicians at the department, who will be acquainted to the study. Results will be collected and checked at the end of the study.

Expected outcomes of the study It's expected that patients in the FG will earn more comfort and regain earlier ROM and strength with no statistically significant differences in complication rate (particularly re-rupture rate) and possible benefits in the end functional outcome.

Dissemination of results and publication policy Publication of the results could bring the support and more confidence in the use of modified percutaneous Achilles tendon repair under local anesthesia with early functional treatment. It could be thus assessed as an effective one (with no more complications and with low costs) and as the method that brings more comfort to the patients with earlier ROM, strength and ability to return to the previous activities in comparison to the concept of rigid postoperative immobilization.

Duration of the project It's designed as a 4-year study.

Problems anticipated Potentially low number of patients who fulfil the inclusion criteria and who will accept to participate in the study, possible problems with the fear in patients of weakness of the functional immobilization, that can be so simply removed, potential problems in respecting the rehabilitation protocol, potential loss of the patients to the final follow-up and potential rejection of the patients to wear rigid immobilization, once they will hear about the comfort and benefits of functional bracing in the patients in the FG (this is one of the reasons for a relatively short duration of the project).

Project management The project will be lead by the main investigator and helped with the co-investigator - all the other employees at the department will be acquainted with the study.

Ethics Presented research will be performed in accordance with the Declaration of Helsinki. The protocol will be considered and approved by the national ethics committee (KME) and will follow ethical standards.

All the patients will be given informed/consent protocol with a free will to take a participation or to decide to any other type of treatment (non-operative or open operative treatment) with a clear presentation of benefits and drawback of each method.

Budget and other support for the project No extra funds will be requested or provided.

Collaboration with other scientists or research institutions No other research institutions will be included.

Links to other projects No link to other projects or groups of investigators.

Other research activities of the investigators Investigators are a full time employees for a clinical work in a state-owned hospital as Orthopaedic-Trauma surgeons.

ELIGIBILITY:
Inclusion Criteria:

* patients 18 years of age or older
* a rupture that occurred no more than 7 days before the operating procedure
* closed, complete ATR
* a rupture that occurred in the tendinous portion (2-8 cm proximal to the insertion)
* informed consent

Exclusion Criteria:

* no previous operative procedures or history of partial or complete rupture of the involved tendon
* no previous local, oral or parenteral therapy that might have weakened the tendon (for instance local infiltration of anesthetics or steroids in the AT region, oral or parenteral immunosuppressive therapy in patients with transplanted organs or immune diseases etc.).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2001-01-01 (Actual); Primary Completion 2004-12-31 (Actual); Study Completion 2007-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Post-operative range of motion | After 2 months, 3 months, 6 months, 12 months and after 3 years post op.
  Assessment in change of dorsiflexion (maximum 0-20 degrees) and plantar flexion (maximum 0-50 degrees), measured with goniometer (Reference: Ryf C, Weyman A. The Neutral Zero Method - A Principle of Measuring Joint Function. Injury. 1995;26(Suppl 1)).
Change in Post-operative strength | After 3 months, 6 months, 12 months and after 3 years post op.
  Heel rise test (rising on toes with both legs, operated leg and non-operated leg, 25 times in 60 seconds). (Reference: Lunsford BR, Perry J. The standing heel-rise test for ankle plantar flexion: criterion for normal. Phys Ther. 1995;75:694-8).
Number of complications | Final results after 3 years
  Clinical findings of occurence
  * Major complications (Rerupture, Second rerupture, Permanent equinus position of the foot, Extreme lengthening of the Achilles tendon, Deep infection, Chronic fistula, Necrosis of the skin, Deep vein Thrombosis, Embolism, Death) and
  * Minor complications (Superficial infection, Wound hematoma, Delayed wound healing, Adhesion of the scar, Disturbances of sensibility, Suture granuloma, Suture rupture)
American Foot and Ankle Society (AOFAS) hindfoot-ankle score | Final result after 3 years
  Filling of AOFAS questionnaire (0 - worst outcome, 100 - best outcome) (reference: 1.Kitaoka HB, Alexander IJ, Adelaar RS, Nunley JA, Myerson MS, Sanders M. Clinical rating systems for the ankle-hindfoot, midfoot, hallux, and lesser toes. Foot Ankle Int. 1994;15:349-53.)

SECONDARY OUTCOMES:
Patient's subjective assessment of treatment | Final assessment after 3 years
  Patient's report: (good) (fair) (poor)
Patient's report to previous activities | Final assessment after 3 years
  Parameters: (no limitation) (with complaints) (not possible)
Patient's report about return to sports activities | Final assessment after 3 years
  Parameters: (no limitation) (with limitations) (not possible)

CONTACTS AND LOCATIONS:
Overall Officials: Andrej Cretnik, MD, PhD, Principal Investigator — University Medical Center Maribor, Ljubljanska 5, 2000 Maribor, Slovenia; Roman Košir, MD, PhD, Principal Investigator — University Medical Center Maribor, Ljubljanska 5, 2000 Maribor, Slovenia
Locations (1):
- University Medical Centre Maribor, Ljubljanska 5, Maribor, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cretnik A, Zlajpah L, Smrkolj V, Kosanovic M. The strength of percutaneous methods of repair of the Achilles tendon: a biomechanical study. Med Sci Sports Exerc. 2000 Jan;32(1):16-20. doi: 10.1097/00005768-200001000-00004. PMID 10647524
- [Background] Wong J, Barrass V, Maffulli N. Quantitative review of operative and nonoperative management of achilles tendon ruptures. Am J Sports Med. 2002 Jul-Aug;30(4):565-75. doi: 10.1177/03635465020300041701. PMID 12130412
- [Background] Cretnik A, Kosanovic M, Smrkolj V. Percutaneous suturing of the ruptured Achilles tendon under local anesthesia. J Foot Ankle Surg. 2004 Mar-Apr;43(2):72-81. doi: 10.1053/j.jfas.2004.01.008. PMID 15057852